CLINICAL TRIAL: NCT00885430
Title: Pico-Salax Colonic Preparation Study: Quantifying Electrolyte and Volume Status Changes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Dr. Lawrence Hookey, Principal Investigator, Queen's University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Hookey Pico-Salax Volunteers
Record Dates: First submitted 2009-04-20; First posted 2009-04-22 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Hemodynamics; Hyponatremia
Keywords: colonoscopy; preparation
MeSH Terms: conditions — Hyponatremia | interventions — Pico-Salax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pico-Salax (Experimental)
  Interventions: Drug: Pico-Salax

INTERVENTIONS:
Drug: Pico-Salax — Two sachets of Pico-Salax given 5 hours apart

SUMMARY:
Twenty adult volunteers will be administered Pico-Salax in the usual fashion for colonoscopy with intense monitoring of serum and urine chemistry and hemodynamics.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers older than 45

Exclusion Criteria:

* impaired renal function
* congestive heart failure ascites known electrolyte abnormalities

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-07; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
serum electrolytes | 48 hours
patient hemodynamics | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Hookey, MD, Principal Investigator — Queen's University
Locations (1):
- Hotel Dieu Hospital, Kingston, Ontario, Canada